CLINICAL TRIAL: NCT02347137
Title: Efficacy of Isolated Whey and Micellar Whey Protein (+/-Citrulline) to Stimulate Protein Synthesis in 'Healthy' and 'Anabolically Resistant' Elderly Muscle
Brief Title: Influence of Reduced Daily Step Count and Anabolic Interventions on Muscle Protein Metabolism in Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11-267
Record Dates: First submitted 2015-01-06; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Older Adults; Muscle Protein Synthetic Response to Protein; Reduced Physical Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isolated Whey Protein (Active Comparator): 20 g isolated whey protein + 15 g non-essential amino acids
  Interventions: Other: step-reduction; Other: step-reduction plus resistance exercise
- Micellar Whey Protein (Experimental): 20 g micellar whey protein + 15 g non-essential amino acids
  Interventions: Other: step-reduction; Other: step-reduction plus resistance exercise
- Micellar Whey Protein + Citrulline (Experimental): 20 g micellar whey protein + 5 g citrulline
  Interventions: Other: step-reduction; Other: step-reduction plus resistance exercise

INTERVENTIONS:
Other: step-reduction — reduce daily physical activity to less than 1500 steps per day
Other: step-reduction plus resistance exercise — reduce physical activity to less than 1500 steps per day with thrice weekly low-load, high effort resistance exercise

SUMMARY:
As the loss of muscle mass with aging is associated with a dysregulation of muscle protein synthesis (MPS) that is generally characterized by an 'anabolic resistance' to nutrients, the primary outcome of the trial is to investigate the effect of a mixed macronutrient beverage on post-prandial myofibrillar MPS. However, the 'anabolic resistance' of aging may be predominantly influenced by the contractile activity of skeletal muscle; for example, the investigators have demonstrated that 2 weeks of reduced habitual activity (i.e. daily step count) induces anabolic resistance in otherwise healthy older adults. In contrast, resistance exercise is well-known to enhance muscle mass and can increase the sensitivity of skeletal muscle to dietary amino acids. Therefore, all participants will undergo a 2-week reduced step count intervention combined with a unilateral leg resistance exercise protocol to induce an 'unhealthy' or 'anabolically resistant' leg and a relatively 'healthy' or 'anabolically sensitive' leg, respectively; this within subject model will be utilized to investigate the effect of the mixed macronutrient beverage in both relatively 'healthy' and 'unhealthy' older muscle. The investigators will also measure changes in muscle mass, muscle function, and cardiovascular health of both legs before and after the 2-week intervention to determine the effect of reduced activity and the protective effect of minimal, low-intensity exercise on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker

Exclusion Criteria:

* Health problems such as: heart disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled hypertension, or any health conditions that might put the participant at risk for this study
* Failed clearance for exercise participation by the participants family physician/medical doctor
* Failed an exercise strength test.
* Regular consumption of any analgesic or anti-inflammatory drug(s), prescription or non-prescription, chronically will be excluded.
* Taking any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Factors that may exclude a participant from an MRI scan (i.e. various implants, metal in the eyes etc)
* Participants who complete fewer than 5000 steps per day (as assessed by pedometer prior to the study).

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Myofibrillar fractional synthetic rate will be measured using 13C6 ring phenylalanine | 7 hours
  analysis

SECONDARY OUTCOMES:
body composition (lean body mass, fat mass, leg lean mass, leg fat mass) will be measured using dual energy xray absorptiometry | 14 days
  analysis
leg muscle strength (leg press and leg extension 1 repetition maximum [1-RM], peak knee extensor torque) will be measured using a dynamometer | 14 days
  analysis
vascular function (femoral blood flow, femoral artery diameter, leg pulse) will be measured using doppler ultrasound | 14 days
  analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Breen L, Stokes KA, Churchward-Venne TA, Moore DR, Baker SK, Smith K, Atherton PJ, Phillips SM. Two weeks of reduced activity decreases leg lean mass and induces "anabolic resistance" of myofibrillar protein synthesis in healthy elderly. J Clin Endocrinol Metab. 2013 Jun;98(6):2604-12. doi: 10.1210/jc.2013-1502. Epub 2013 Apr 15. PMID 23589526
- [Background] Burd NA, West DW, Moore DR, Atherton PJ, Staples AW, Prior T, Tang JE, Rennie MJ, Baker SK, Phillips SM. Enhanced amino acid sensitivity of myofibrillar protein synthesis persists for up to 24 h after resistance exercise in young men. J Nutr. 2011 Apr 1;141(4):568-73. doi: 10.3945/jn.110.135038. Epub 2011 Feb 2. PMID 21289204